CLINICAL TRIAL: NCT04474002
Title: Efficacy, Tolerance and Safety of Split Dose Bowel Preparation for Colonoscopy: 4L Polyethylene Glycol (PEG) Versus 1L Polyethylene Glycol Plus Sodium Picosulfate-magnesium Citrate (SPMC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Tso Yau Kan, Resident, Queen Elizabeth Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PICO-PEG trial
Record Dates: First submitted 2020-07-12; First posted 2020-07-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Bowel Preparation Solutions; Colonoscopy
Keywords: Polyethylene glycol; Picoprep; Cathartics; Bowel preparation solution; Colonoscopy
MeSH Terms: interventions — klean prep

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4L Klean Prep® (Active Comparator): Drug: 59g polyethylene glycol, 5.685g Na sulphate, 1.685g Na bicarbonate, 1.465g NaCl, 0.7425g KCl and aspartame 0.0494g
  Interventions: Drug: 4L Klean Prep®
- 1L Klean prep® and 2 sachets Picoprep® (Experimental): Drug: 59g polyethylene glycol, 5.685g Na sulphate, 1.685g Na bicarbonate, 1.465g NaCl, 0.7425g KCl, aspartame 0.0494g, sodium picosulfate 0.01g, magnesium oxide 3.5g, citric acid 12.0g
  Interventions: Drug: 1L Klean prep® and 2 sachets Picoprep®

INTERVENTIONS:
Drug: 4L Klean Prep® — Patients allocated to the control group shall mix two sachets of PEG in 2L water. At 6pm the evening before examination, they shall consume 250ml solution every 15mins, and finish in 2hours. At 7am the day of examination, drink another 2L Klean-prep in 2 hours.
  Arms: 4L Klean Prep®
Drug: 1L Klean prep® and 2 sachets Picoprep® — Patients allocated to the study group shall mix each sachet of Picoprep® in 150ml warm water. The patient shall take the 1st dose at 4pm the day before procedure followed by at least five 250ml drinks of clear fluid before the next dose. The 2nd dose shall be taken approximately 6hrs later and followed by at least three 250ml drinks of clear fluid before bed. On 7am the day of procedure, they shall take 1L PEG in 1 hour.
  Arms: 1L Klean prep® and 2 sachets Picoprep®

SUMMARY:
4L split dose PEG is the gold standard for bowel preparation, however it comes with poor tolerability and poor compliance. Combination of PEG with different agent is useful in reducing total volume, improving compliance and tolerance of patient.

The objective of this study is to demonstrate that combination bowel preparation, PEG plus SPMC solution, has similar efficacy and safety profile whereas with a better tolerance when compared to large volume PEG.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-center, single-blinded, non-inferiority trial.

Participants with out patient colonoscopy arranged will be included and randomized in a 1:1 ratio to receive either a split dose of 4L PEG + Electrolyte (Klean-prep® ) or 1L Klean-prep® plus 2 sachets SPMC (Picoprep®).

Trained endoscopists will be using the Boston Bowel Preparation Scale (BBPS) to assess the quality of bowel preparation. Patient would also rate the tolerance, compliance and adverse effect by filling the questionnaire before the colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who mentally capable to consent for participating the trial
2. 18 - 65 years old
3. Scheduled for 1st colonoscopy
4. Elective outpatient colonoscopy

Exclusion Criteria:

1. Prior colorectal or abdominal-pelvic surgery
2. Inflammatory bowel disease
3. Active bowel condition eg intestinal obstruction
4. Gastrointestinal disorders eg active ulcer, gastric outlet obstruction, gastroparesis and hypomotility syndrome
5. Recent myocardial infarction, congestive heart failure, uncontrolled hypertension
6. Renal dysfunction, hepatic disease
7. Patient on long term tranquilizer, anti-spasmodic, prokinetic, laxative or antidiarrhoeal agents
8. Hypersensitivity to PEG or SPMC solution
9. Pregnant or breastfeeding women
10. Inability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Score (BBPS) | Up to 24 weeks
  Adequate bowel preparation is defined as a total BPPS score >/= 6 in which all three segments had score >/=2

SECONDARY OUTCOMES:
Patient tolerability to bowel preparation using Likert scale | Up to 24 weeks
  Patient are requested to fill in questionnaire on the day of colonoscopy. Candidate are asked to rate the frequency of complications between 'none', 'mild', 'moderate' and 'severe'. 'None' being the best outcome and 'severe' being the worst outcome.
Patient compliance towards bowel preparation | Till the day of procedure
  Proportion of patient able to complete the whole bowel preparation as instructed by protocol
Proportion of patient requiring repeat colonoscopy | Up to 24 weeks
  Proportion of incomplete colonoscopy due to inadequate bowel preparation Patient will be attended by physicians and blood taking will be arranged
Incidence of treatment related adverse events | Up to 24 weeks
  Patient will be monitored after colonoscopy for any complications

CONTACTS AND LOCATIONS:
Overall Officials: Yau Kan Tso, Principal Investigator — Queen Elizabeth Hospital, Hospital Authority
Locations (1):
- Queen Elizabeth Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT04474002/ICF_000.pdf